CLINICAL TRIAL: NCT03529149
Title: TCD Monitoring Technology Guides the Precise Control of Blood Pressure After EVT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: [2018]007
Record Dates: First submitted 2018-04-22; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — urapidil; Diltiazem; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Accurate blood pressure control (Experimental): Implementing accurate blood pressure management under TCD monitoring
  Interventions: Combination Product: Urapidil Hydrochloride Injection
- Guideline blood pressure control (Active Comparator): Control blood pressure according to guidelines
  Interventions: Combination Product: Urapidil Hydrochloride Injection

INTERVENTIONS:
Combination Product: Urapidil Hydrochloride Injection — Accurate monitoring of blood pressure is carried out under TCD monitoring, that is to maintain （mean flow velocity）MFV or （pulse index）PI target blood pressure. The target values of MFV and PI are MFV>37cm/s of （middle cerebral artery)MCA, PI < 1.34cm/s, aMFV>40cm/s of (basilar artery)BA, PI < 0.8cm/s.
  TCD shows that when the MFV of MCA or BA is lower than the target value, the blood pressure is reduced or discontinued according to the insufficiency of blood flow. and the current blood pressure is maintained once MFV is met. TCD showed that the PI index of MCA or BA was higher than the target value . The blood pressure reduction was treated by excessive perfusion: intravenous infusion of blood pressure drugs , once PI index is up to the standard, maintaining the current blood pressure.
  Other Names: Diltiazem Hydrochloride for Injection

SUMMARY:
Investigators hypothesized that the precise regulation of blood pressure based on the changes of cerebral blood flow parameters under TCD monitoring can better improve the state of cerebral blood flow, reduce the risk of early neurological deterioration and improve the prognosis of the patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* accept EVT treatment within 6 hours of symptoms onset;
* In selected patients with AIS within 6 to 16 hours of last known normal who have LVO in the anterior circulation and meet other DAWN or DEFUSE 3 eligibility criteria..
* In selected patients with AIS within 6 to 24 hours of last known normal who have LVO in the anterior circulation and meet other DAWN eligibility criteria.

Exclusion Criteria:

* Pre - onset mRS>2;
* severe dementia;
* threatening life diseases (such as malignant tumor, etc.);
* non acute ischemic cerebrovascular disease patients undergoing selective intravascular treatment;
* related sound window closure can not be monitoring with TCD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-04-08 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
early neurological deterioration | 72 hours
  the incidence of 72 hours in National Institute of Health stroke scale increased more than 4 points or National Institute of Health stroke scale Ia score more than 1 points

SECONDARY OUTCOMES:
prognosis of nerve function | 3 months
  prognosis of nerve function use Modified Rankin Scale,0~3 is good prognosis and 4~6 is poor prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No